CLINICAL TRIAL: NCT04659408
Title: The Effect of Probiotic and Prebiotic Supplementation on Gastrointestinal Comfort in Elite Athletes with Spinal Cord Injury: a Pilot Study
Brief Title: Probiotic and Prebiotic Supplementation in Elite Athletes with Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2020-03
Record Dates: First submitted 2020-11-24; First posted 2020-12-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2021-12

CONDITIONS: Spinal Cord Injuries
Keywords: probiotic supplementation; prebiotic supplementation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with within-participants crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bactosan - oat bran (Experimental): This group will receive Bactosan first, followed by oat bran.
  Interventions: Dietary Supplement: Multistrain probiotic preparation; Dietary Supplement: Oat Bran
- Oat bran - Bactosan (Experimental): This group will receive oat bran first, followed by Bactosan.
  Interventions: Dietary Supplement: Multistrain probiotic preparation; Dietary Supplement: Oat Bran

INTERVENTIONS:
Dietary Supplement: Multistrain probiotic preparation — One sachet daily, containing 3 grams of the freeze-dried multispecies probiotic Bactosan for a period of four weeks. One sachet will be mixed with 50-100 ml water and taken daily before breakfast or dinner. Bactosan contains the following eight bacterial strains: Bifidobacterium lactis W51, Bifidobacterium lactis W52, Enterococcus faecium W54, Lactobacillus acidophilus W22, Lactobacillus paracasei W20, Lactobacillus plantarum W21, Lactobacillus salivarius W24 and Lactococcus lactis W19, with a total viable cell count of 1 × 109 cfu/gram, and therefore 3 × 109 cfu/daily dose.
  Other Names: BactoSan pro FOS (Mepha, Switzerland)
Dietary Supplement: Oat Bran — 5 grams (one teaspoon) daily of the oat bran together with a meal of preference. The oat bran can be added to the usual breakfast cereal, yoghurt, pancakes, juice, milk, salad sauce or in an omelette.
  Other Names: Naturaplan Organic Oat Bran (Coop, Switzerland)

SUMMARY:
The main objective of this pilot study is to obtain information, which will be used for the design of a main randomized controlled trial (RCT) with a larger size based on feasibility, validity and sample size estimation as well as the potential effects of pre- and probiotic intake on intestinal microbiota. A larger trial will then be designed to test the hypothesis that adding probiotics or prebiotics may improve gut microbiome composition, gastrointestinal symptoms as well as cardiometabolic health indices in mid-term and possibly lead to improved sports performance over a longer-term period in athletes with a Spinal Cord Injury.

DETAILED DESCRIPTION:
In this pilot crossover randomized controlled trial, twenty (N = 20) para-athletes will participate in an intervention consisting of a four-week intake of probiotic, using the commercially available multistrain probiotic preparation "BactoSan pro FOS" from Mepha (Basel, Switzerland), followed by a four-week wash-out period, and a four-week prebiotic intervention using "Naturaplan Bio Oat Bran" (Coop, Switzerland). Total duration of the study will be 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* athletes with a spinal cord injury shortlisted as potential participants for major international events, such as the Paralympic Games 2021 in Tokyo and World Championship qualification

Exclusion Criteria:

* Chronic inflammatory bowel diseases (i.e. ulcerative colitis, Crohn's disease)
* Taking antibiotics and/or other medication to alleviate gastrointestinal complaints at recruitment time point
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | At baseline
  Proportion of invited participants who agreed to participate in the trial
Dropout rate | Through study completion, an average of 4 months
  The proportion of randomized participants who did not complete the study protocol
Severe adverse events | Through study completion, an average of 4 months
  The occurrence of severe adverse events (SAEs)

SECONDARY OUTCOMES:
Gastrointestinal problems | At 0, 1, 2, 3 months
  Assessed using the Gastrointestinal Quality of Life Index (GIQLI) of Eypasch, using a 5-point scale (0-4) with total range 0-144 and higher scores indicating better outcomes.
Stool microbiome characterization | At 0, 1, 2, 3 months
  Stool probes will be sampled by the participants at home and send to the study center. The "What's in my Pot?" (WIMP) workflow (Oxford Nanopore Technologies) will be used to classify and identify species in real time, generating a graphical WIMP report of the sample composition and the most reliable placement in the taxonomy tree, assigning a score to each taxonomic placement.
Monitoring of inflammation | At 0, 1, 2, 3 months
  C-reactive protein (CRP) from blood samples in mg/L
Loss of training days due to injury or illness | At 0, 1, 2, 3 months
  Assessed using the Oslo Sports Trauma Research Centre (OSTRC) Overuse Injury Questionnaire, which consists of several multiple choice and open questions (no scale).
Food intake during three days | At 0, 1, 2, 3 months
  Self-reported intake (content and quantity) of food on a data sheet, including photo's. Calculations of the nutritional quality and quantity of consumed foods, drinks and nutritional supplements will be performed using PRODI® Swiss, a computer program for nutritional counselling and nutritional therapy.
Recording of leisure time activity | At 0, 1, 2, 3 months
  Assessed using the Leisure Time Physical Activity Questionnaire (LTPA-Q), which records number of days and minutes of physical activity (no scale).

CONTACTS AND LOCATIONS:
Overall Officials: Joëlle Flück, PhD, Principal Investigator — Sports nutrition expert
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hertig-Godeschalk A, Glisic M, Ruettimann B, Valido E, Capossela S, Stoyanov J, Flueck JL. The feasibility of a randomized controlled crossover trial to assess the effect of probiotic and prebiotic supplementation on the health of elite wheelchair athletes. Pilot Feasibility Stud. 2023 Jun 15;9(1):99. doi: 10.1186/s40814-023-01339-6. PMID 37322538
- [Derived] Glisic M, Flueck JL, Ruettimann B, Hertig-Godeschalk A, Valido E, Bertolo A, Stucki G, Stoyanov J. The feasibility of a crossover, randomized controlled trial design to assess the effect of probiotics and prebiotics on health of elite Swiss para-athletes: a study protocol. Pilot Feasibility Stud. 2022 Apr 27;8(1):94. doi: 10.1186/s40814-022-01048-6. PMID 35477496